CLINICAL TRIAL: NCT06108336
Title: Investigation of Cerebellar Involvement in Cognitive Sequencing
Brief Title: Cerebellar Involvement in Cognitive Sequencing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00328214; R01MH128278 (NIH)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Effects of Cerebellar Stimulation on Brain Activation
Keywords: sequencing; cerebellum; transcranial magnetic stimulation; TMS; functional MRI; fMRI; verbal working memory
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Cerebellar and Occipital stimulation groups will be tested under sequence-demanding and non-sequence demanding tasks (in counterbalanced order)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebellar Stimulation (Experimental): TMS will be administered to the cerebellum on half the trials of a sequence-demanding task, and on half the trials of a non-sequence-demanding task. Task order will be counterbalanced.
  Interventions: Procedure: TMS during sequence-demanding task; Procedure: No TMS during sequence-demanding task; Procedure: TMS during non-sequence-demanding task; Procedure: No TMS during non-sequence-demanding task
- Occipital Stimulation (Active Comparator): TMS will be administered to an occipital control region on half the trials of a sequence-demanding task, and on half the trials of a non-sequence-demanding task. Task order will be counterbalanced.
  Interventions: Procedure: TMS during sequence-demanding task; Procedure: No TMS during sequence-demanding task; Procedure: TMS during non-sequence-demanding task; Procedure: No TMS during non-sequence-demanding task

INTERVENTIONS:
Procedure: TMS during sequence-demanding task — TMS is administered during the execution of sequence-demanding task. Transcranial magnetic stimulation (TMS) is a safe and non-invasive technique for transiently modulating brain activity
  Other Names: Transcranial magnetic stimulation
Procedure: No TMS during sequence-demanding task — TMS is not administered during the execution of sequence-demanding task.
Procedure: TMS during non-sequence-demanding task — TMS is administered during the execution of non-sequence-demanding task. Transcranial magnetic stimulation (TMS) is a safe and non-invasive technique for transiently modulating brain activity
Procedure: No TMS during non-sequence-demanding task — TMS is not administered during the execution of non-sequence-demanding task

SUMMARY:
Although there is increasing recognition that the cerebellum is involved in cognition as well as motor function, the manner in which the cerebellum contributes to cognition is uncertain. One theory that might account for both motor and cognitive contributions of the cerebellum is that the cerebellum is involved in sequencing of relevant events or stimuli. Previous experiments have suggested that disruption of the cerebellum impairs the prediction of the next event in a sequence. The present experiment will examine the impact of cerebellar stimulation on brain activation during the performance of both sequence-demanding and non-sequence-demanding tasks.

DETAILED DESCRIPTION:
Although there is increasing recognition that the cerebellum, which contains half of the brain's neurons, is involved in cognition as well as motor function, the manner in which the cerebellum contributes to cognition is uncertain. The uniform circuitry of the cerebellum and the extensive connectivity of the cerebellum with numerous neocortical regions has suggested to some researchers that there is a common computation that the cerebellum performs for both motor and cognitive functions. The cerebellar sequencing hypothesis posits that the cerebellum acquires sequence information, makes sequence predictions, and detects sequence violations. These functions, executed via a forward model, could underlie cerebellar involvement in both motor and cognitive behavior. In motor control, such predictions can be used to guide limb trajectory without reliance on movement-generated sensory feedback. In cognition, sequencing requirements are prominent in both verbal working memory (VWM) and language acquisition; eg, in VWM, keeping a phone number in mind requires encoding and rehearsing a sequence of digits. In language, words consist of sequences of syllables, and the learning of syllable transition probabilities is an important component of recognizing legal words in a language. Importantly, prominent cerebellar activation has been observed in many functional MRI (fMRI) VWM and language studies. However, the brainstem/cerebellar neural correlates of sequencing in cognition, and the influence of cerebellar sequence predictions on neocortical targets, are poorly understood. In this experiment, studying healthy individuals the investigators will Investigate the cerebellum as a source of sequence prediction and its influence on forebrain areas. The cerebellum is hypothesized to provide its forward model sequence prediction to forebrain targets, but to date no study has attempted to visualize with concurrent TMS/fMRI the consequences of disrupting this cerebellar input on forebrain activation. In the investigators previous work, the investigators show that transcranial magnetic stimulation (TMS) during the rehearsal of a sequence of letters results in errors in determining if a probe letter matches the next letter in the sequence, suggesting that TMS disrupted this predictive input. In accordance with this finding, the investigators hypothesize that, using concurrent TMS/fMRI, TMS disruption during a sequencing task will produce greater changes in neocortical activation relative to an analogous control task that does not have the predictive component brought out by sequencing demands. The investigators further hypothesize that different patterns of neocortical activations in response to cerebellar TMS will be observed depending on whether a probe letter matches the expected next letter in a sequence.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-50;
* 2) educational attainment of at least 8 years;
* 3) capable of giving informed consent;
* 4) fluent speaker of English by self-report;
* 5) right handed.

Exclusion Criteria:

* 1) illicit drug use within 30 days of MRI scanning;
* 2) neurological or systemic disorder which can cause dementia or cognitive dysfunction;
* 3) history of an Axis I psychiatric disorder including substance use disorder;
* 4) history of definite stroke;
* 5) focal lesion on MRI exam;
* 6) uncorrected visual deficits by self-report
* 7) contraindications for MRI scanning
* 8) use of anxiolytic, antidepressant, neuroleptic, or sedative medication
* 9) Additional exclusion criteria recommended by Wassermann for TMS neuromodulation, including: History of seizure or a family history of epilepsy, heart disease, intracardiac lines, increased intracranial pressure, history of head trauma, and history of respiratory disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
functional magnetic resonance imaging brain activation | during scan up to 1 hour
  functional magnetic resonance imaging brain activation. For the sequential task, a sequence of letters is presented and the subject is presented with number signs, one at a time, to guide rehearsal of the sequence. At some point a probe letter is presented and the subject indicates by button press if the probe is the next letter in the sequence. For the non-sequential task, subjects do not have a guided rehearsal, and the response to the probe indicates if the probe was one of the letters originally presented. Brain activation in response to the probe will be measured with brain stimulation vs no brain stimulation for each task

SECONDARY OUTCOMES:
percent correct of behavioral responses | during scan up to 1 hour
  percent correct of behavioral responses. For the sequential task, a sequence of letters is presented and the subject is presented with # signs, one at a time, to guide rehearsal of the sequence. At some point a probe letter is presented and the subject indicates by button press if the probe is the next letter in the sequence. For the non-sequential task, subjects do not have a guided rehearsal, and the response to the probe indicates if the probe was one of the letters originally presented. Behavioral accuracy consists of the percent of correct responses to the probe, with higher numbers indicating better performance
behavioral reaction time (milliseconds) | during scan up to 1 hour
  behavioral reaction time to respond to the probe. Increases in reaction time indicate greater difficulty for the subject to respond

CONTACTS AND LOCATIONS:
Overall Officials: John E Desmond, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States